CLINICAL TRIAL: NCT00776776
Title: Follow-up of Adolescent Bariatric Surgery
Acronym: FABS
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Thomas H. Inge, MD, PhD, Principal Investigator, Cincinnati Children's Hospital Medical Center
Other Study IDs: 2008-0954
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2008-08

CONDITIONS: Morbid Obesity
Keywords: BMI > 40; Obesity; Adolescents; Weight Loss Surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Very little information is available about extremely obese (body mass index [BMI] > 40 kg/m2) adolescents. The purpose of the Follow up of Adolescent Bariatric Surgery (FABS) study is to collect information obtained during the clinical care of obese adolescents from all over the country that can be used by researchers to study obesity, the complications of obesity, and the outcomes of obesity treatment during adolescence. This information will be used to describe the experience of the obese adolescent, including how obesity during adolescence and its treatment impacts health and well-being. The information may also be used to study causes of obesity, to determine the predictors of successful obesity treatment and for other obesity related research. Because of the importance of understanding the outcome of obesity and obesity treatments (surgical and non-surgical) on the patient over time, the data included in the study will be collected before, during and after any treatments rendered. For those who do not undergo a treatment which results in major weight change, it will be critical to determine the natural history of adolescent severe obesity as the adolescent transitions into adulthood. Finally, another important purpose of the FABS research study is to obtain patients' consent to be contacted for possible participation in future research studies.

SPECIFIC AIMS:

1. To describe the natural history of morbid obesity among adolescents who seek treatment for their obesity
2. To describe major outcomes following bariatric surgery in adolescents evaluated at 3, 6, 12, and annually for 10 years post-operatively and compare these to outcomes to patients managed non-surgically
3. To organize a national cohort of severely obese adolescents who agree to be contacted in the future for research studies

ELIGIBILITY:
Inclusion Criteria:

* All patients seeking treatment for Obesity at Cincinnati

Exclusion Criteria:

* Currently Enrolled in Teen LABS Study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients Seeking Treatment for Obesity at Cincinnati Children's Hosptial Medical Center in Cincinnati, OH.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
BMI | Annually

SECONDARY OUTCOMES:
Medical Co-morbidities | Annual

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Kalra M, Inge T, Garcia V, Daniels S, Lawson L, Curti R, Cohen A, Amin R. Obstructive sleep apnea in extremely overweight adolescents undergoing bariatric surgery. Obes Res. 2005 Jul;13(7):1175-9. doi: 10.1038/oby.2005.139. PMID 16076986
- [Result] Xanthakos SA, Inge TH. Nutritional consequences of bariatric surgery. Curr Opin Clin Nutr Metab Care. 2006 Jul;9(4):489-96. doi: 10.1097/01.mco.0000232913.07355.cf. PMID 16778582
- [Result] Miller RJ, Xanthakos SA, Hillard PJ, Inge TH. Bariatric surgery and adolescent gynecology. Curr Opin Obstet Gynecol. 2007 Oct;19(5):427-33. doi: 10.1097/GCO.0b013e3282efb285. PMID 17885457
- [Result] Roehrig HR, Xanthakos SA, Sweeney J, Zeller MH, Inge TH. Pregnancy after gastric bypass surgery in adolescents. Obes Surg. 2007 Jul;17(7):873-7. doi: 10.1007/s11695-007-9162-7. PMID 17894144
- [Result] Ippisch HM, Inge TH, Daniels SR, Wang B, Khoury PR, Witt SA, Glascock BJ, Garcia VF, Kimball TR. Reversibility of cardiac abnormalities in morbidly obese adolescents. J Am Coll Cardiol. 2008 Apr 8;51(14):1342-8. doi: 10.1016/j.jacc.2007.12.029. PMID 18387434
- [Derived] Inge TH, Jenkins TM, Xanthakos SA, Dixon JB, Daniels SR, Zeller MH, Helmrath MA. Long-term outcomes of bariatric surgery in adolescents with severe obesity (FABS-5+): a prospective follow-up analysis. Lancet Diabetes Endocrinol. 2017 Mar;5(3):165-173. doi: 10.1016/S2213-8587(16)30315-1. Epub 2017 Jan 6. PMID 28065736